CLINICAL TRIAL: NCT00153582
Title: Phase II Study of WT1 126-134 Peptide Vaccination in Combination With Adjuvants GM-CSF and KLH in AML
Brief Title: WT1 Peptide Vaccination in Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaemaCBFWT102; Carreras 04/25f
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2005-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

INTERVENTIONS:
Biological: WT1 126-134 peptide

SUMMARY:
In this trial, HLA-A2+ patients with active AML are vaccinated with a peptide from the leukemia-associated antigen WT1 together with immunological adjuvants keyhole limpet hemocyanin (KLH) as T-helper protein and granulocyte macrophage colony stimulating factor (GM-CSF) 4 times bi-weekly, then monthly.

DETAILED DESCRIPTION:
In this phase II trial HLA-A2+ patients with active AML without curative treatment option are vaccinated with WT1 126-134 peptide mixed with adjuvant KLH as T-helper protein and GM-CSF 4 times bi-weekly, then monthly.

ELIGIBILITY:
Inclusion Criteria:

* AML or myelodysplastic syndromes (MDS)
* Partial response (PR) or complete response (CR) or smoldering course without option for allogeneic stem cell transplantation
* HLA-A2+
* WT1-expression in bone marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2002-04

PRIMARY OUTCOMES:
Generation of T cell response

SECONDARY OUTCOMES:
Clinical outcome
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité
Locations (1):
- Hematology&Oncology Charité CBF, Berlin, Germany

REFERENCES:
- [Result] Mailander V, Scheibenbogen C, Thiel E, Letsch A, Blau IW, Keilholz U. Complete remission in a patient with recurrent acute myeloid leukemia induced by vaccination with WT1 peptide in the absence of hematological or renal toxicity. Leukemia. 2004 Jan;18(1):165-6. doi: 10.1038/sj.leu.2403186. No abstract available. PMID 14603333